CLINICAL TRIAL: NCT04490330
Title: Screening for Alcohol-related Cognitive Impairments in Cirrhotic Patients
Acronym: CirCo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0106
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Alcohol Dependence; Dependence; Cognitive Impairments; Cirrhosis; Liver Diseases
Keywords: Alcohol Dependence; Dependence; Cognitive Impairments; Cirrhosis; Liver Diseases
MeSH Terms: conditions — Alcoholism; Cognitive Dysfunction; Fibrosis; Liver Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — AUDIT questionnaire (alcohol use disorders identification test)

SUMMARY:
80% of patients with alcohol use disorders (AUD) present cognitive impairments, such as memory and executive functions. These disorders may have repercussions in addiction treatment by altering the patient's adherence to care. The level of impairment is dependent on the onset of addiction, and also the duration of abstinence.

A complete neuropsychological evaluation is necessary to highlight cognitive impairments. In practice, the evaluation of these disorders by practitioners, is done with the help of tools of screening like the MoCa (Montreal cognitive assesment) and the BEARNI (Brief evaluation of alcohol related neuropsychological impairment).

However, none of these tools have been evaluated in patients with alcoholic cirrhosis. Indeed, some studies have suggested that liver disorders including cirrhosis may be a factor aggravating cognitive disorders.

The purpose of this study is to evaluate the ability of the BEARNI tool to detect alcohol-related cognitive problems in patients with alcohol-related cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cirrhosis
* patients with cirrhosis diagnosed by clinical examination
* patients with cirrhosis diagnosed by biological and / or morphological and / or noninvasive tests and / or liver biopsy
* CHILD A, B or C

Exclusion Criteria:

* hepatitis encephalopathy less than 6 months old
* complicated cirrhosis with hepatocellular carcinoma
* Acute alcoholic hepatitis
* viral cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic cirrhosis will be evaluated with BEARNI tool in order to detect alcohol-related cognitive problems.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
number of alcoholic cirrhosis patients with presence of alcohol-related cognitive disorders | day 1
  the number of alcoholic cirrhosis patients with presence of alcohol-related cognitive disorders will be measured by using the BEARNI screening tool. BEARNI screening tool is Brief evaluation of alcohol related neuropsychological impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No